CLINICAL TRIAL: NCT04509349
Title: Alternating Current Stimulation for Essential Tremor: a Pilot Study to Identify the Most Promising Strategy
Brief Title: Alternating Current Stimulation for Essential Tremor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB20-0889
Record Dates: First submitted 2020-07-20; First posted 2020-08-12 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tACS (Active Comparator): For transcranial stimulation, a stimulation method called high-definition tACS (HD-tACS) will be applied to target the primary motor cortex (M1), an area of the brain that is involved in controlling movement, using gel electrodes placed on the scalp. Participant will wear an electrode cap with 5 gel-filled cup HD electrodes arranged in a 4 x 1 montage, to create focused stimulation over the M1 region. A stimulator will be connected to the electrodes to deliver a low-intensity stimulating current to the scalp.
  Interventions: Device: transcranial Altering Current Stimulation; Device: Sham tACS
- Sham tACS (Placebo Comparator): For the transcutaneous ACS, the procedure for real and sham stimulation will be identical to HD-tDCS, but ACS will be delivered to the upper arm contralateral to hand attached to the accelerometer.
  Interventions: Device: transcranial Altering Current Stimulation; Device: Sham tACS

INTERVENTIONS:
Device: transcranial Altering Current Stimulation — The participant will wear an electrode cap with 5 gel-filled cup HD electrodes arranged in a 4 x 1 montage.
Device: Sham tACS — 2 saline sponge electrodes will be attached to the upper arm contralateral to hand attached to the accelerometer.

SUMMARY:
Movement disorders are common neurological disorders, characterized by either excess or paucity of movements. Essential tremor (ET) is one of the most common of these disorders, defined as chronic, rhythmic involuntary movements (tremor) that occur primarily during action involving the upper extremities as prominent body site. ET occurs in between 0.4% and 4% of adults below age 60, its prevalence and related impairment of routine daily actions increasing dramatically with age. More than half of patients do not regain functional independence with medications. These patients are offered functional neurosurgical approaches that carry procedural risk or adverse effects secondary to deep electric stimulation of surgical lesioning. Hence, there is a substantial need for alternative, non-invasive therapeutic options for this disabling neurological disorder. Recently, non-invasive neuromodulation applied as transcranial alternating current stimulation (tACS), has emerged as promising for tremor control. In healthy subjects, tACS applied with a high definition (or focused) montage to the primary motor cortex (M1), was found to entrain physiological tremor; in patients with Parkinson's disease, tACS could decrease the amplitude of rest tremor when the stimulation was delivered in phase with, and at the same frequency of, the tremor. Tremor in ET could also be entrained applying ACS to the arm skin's peripheral nerves (transcutaneous ACS), but its effect on tremor amplitude is unknown.

METHODS AND POTENTIAL CONTRIBUTION/IMPACT OF THE RESEARCH.

The proposed project aims to explore the whole potential of tACS for the tremor suppression in ET. The investigators aim to test the following hypotheses:

1. focused (or high definition, HD) tACS delivered over M1 at the same frequency of the tremor is effective in decreasing tremor amplitude in ET;
2. this effect is strongest when the delivery of tACS is locked to the phase of the tremor expressed by the patient, i.e. administering tACS in a closed-loop modality;
3. transcutaneous ACS in the upper extremities is as effective as tACS applied to the scalp around M1.

DETAILED DESCRIPTION:
This investigation will collect preliminary data on the efficacy of real vs. sham, as well as unlocked vs. phase-locked, modalities of tACS and transcutaneous ACS on tremor amplitude in 25 patients with ET.

Comparing transcranial and transcutaneous, as well as unlocked and phase-locked, modalities represents the novelty of our approach. This has the potential to generate a wealth of preliminary data forming the basis of a large, randomized controlled trial of multiple sessions of this intervention, hence potentially capable of producing long-lasting effects, in this common and disabling disorder. Given its non-invasiveness and relatively low cost, this approach has, if effective, a huge therapeutic potential in ET.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet Diagnostic and Statistical Manual of Mental Disorders criteria for ET (APA, DSM V).
* 18 years of age or older.
* Participants should be either un-medicated or on stable medication treatment for tremor for the previous 3 months.
* Psychiatric comorbidities should be clinically stable; treatment has not changed in the last 3 months.

Exclusion Criteria:

* Have a metal object/implant in their brain, skull, scalp, or neck.
* Have an implantable device (e.g., cardiac pacemaker).
* Have a diagnosis of epilepsy or cardiac disease.
* Have a history of traumatic brain injury, learning disability or dyslexia.
* Have a severe impediment in vision or hearing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Essential Tremor Severity Change | Right before and immediately after the intervention
  The tremor severity will be assessed in the participants by a Movement Disorders Neurologist.

CONTACTS AND LOCATIONS:
Overall Officials: Davide Martino, MD, PhD, Principal Investigator — Department of Clinical Neurosciences, University of Calgary

IPD SHARING:
Plan to Share IPD: No